CLINICAL TRIAL: NCT02492971
Title: Development of a Function-oriented Assistive Technology Indexing System and Its Promotion in the Disabled Population
Brief Title: Function-oriented Assistive Technology Indexing System Development and Promotion
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: kcheng
Record Dates: First submitted 2015-03-16; First posted 2015-07-09 (Estimated); Last update posted 2018-01-25 (Actual); Status verified 2017-11

CONDITIONS: Multiple Disability
Keywords: Assistive technology; functional needs; system usability

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Appropriate assistive devices are important factors for the activity participation of the disabled. These devices should be prescribed by the specialists based on their functional needs. However, most individuals in need of assistive devices locate in the household, school, or nursing institute, in which the professional interventions are not always available on demand. Consequently most assistive devices are used without thorough evaluation, therefore do not necessarily meet the exact needs of the individual. Hence an easy-to-access and easy-to-use assistive technology device indexing system based on the functional needs of the subjects is necessary. The goals of this two-year study are twofold: assistive technology indexing system application(APP) development and promotion. First, the multidisciplinary research team, composed of specialists from assistive technology, rehabilitation, computer science, and special education fields, is going to integrate and refine the current resources and develop an assistive technology indexing system App based on the functional needs of the disabled. Second, in cooperation with the disabled community and special schools, the team is going to promote the use of the App and evaluate its usability via System Usability Scale. This App will be beneficial to the individuals in need of assistive device application. It can also be used as an assistive device manual for the specialists. The App will guide the individuals step by step to the proper assistive devices based on their functional capacities. The complete system will include details of each assistive device and link up with the related service resources. With its registering function, the statistics collected via user clicks can serve as references for further design adjustments and assistive device related policy modifications. All together this App can provide comprehensive services to the disabled in need of assistive devices.

ELIGIBILITY:
Inclusion Criteria:

Caregivers:

1. ages ranged from 20 to 60 years old,
2. serves as the primary caregiver of the disabled in school and organization settings,
3. minimum 6 months caring experience, at least 10 hours direct contact with the client per week.

People with disabilities:

1. ages ranged from 20 to 60 years old,
2. experienced with assistive devices use at least for 1 year,

Exclusion criteria:

* Any visual or motor problems that restrain the use of a smart phone.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: the disabled and their caregivers
Sampling Method: Non-Probability Sample
Enrollment: 175 (Actual)
Dates: Start 2016-09; Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
user satisfaction (by using System Usability Scale) | up to 30 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Hsin-Yi K Kathyju@hotmial.com, phD, Principal Investigator — Chang Gung University
Locations (1):
- Chang Gung Univ., Taoyuan District, Taiwan